CLINICAL TRIAL: NCT02339662
Title: Prospective, Cross Over Gabapentin vs Amitriptyline Study on Patients Suffering From Masticatory Muscle Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Doron Aframian (Other)
Responsible Party: Sponsor-Investigator, Doron Aframian, Professor in Oral Medicine, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: gbvsam001-HMO-CTIL
Record Dates: First submitted 2014-12-14; First posted 2015-01-15 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Myofacial Pain
MeSH Terms: conditions — Facial Pain | interventions — Gabapentin; Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gabapentin (Active Comparator): 900 mg per day total, 3 pills of 300mg.
  Interventions: Drug: Gabapentin
- amitriptyline (Active Comparator): 20 mg total, 1pill
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Gabapentin — muscles pain treatment
  Arms: gabapentin
Drug: Amitriptyline — muscles pain treatment
  Other Names: alterolet
  Arms: amitriptyline

SUMMARY:
The purpose of the study is comparing two drugs efficacy for the treatment of pain originates from masticatory muscles. The two drugs are - Amitriptlyne (amitriptyline) and Gabapentin (gabapentin), both of them are common use in for the treatment of chronic pain Methods - patient that is diagnosed as suffering from myofacial pain, will receive one of the medications above (Gabapentin or amitriptyline) for one month only, after which he will be invited to pain clinic for control. Two weeks after that, the patient will start taking the other drug for 1 month and then invited again to the department for recall and continue standard treatment . The patient can choose whether to continue medication with one of the drugs or stop this medication treatment. Total duration of the experiment is two and a half months.

DETAILED DESCRIPTION:
Temporomandibular disorder is one of the main reasons for the pain and damage to the function in the head, jaws and neck (1,2) term is somewhat misleading because it includes two types of pain, one originates from the temporomandibular joint , and another originates mainly from the muscles of mastication - Myofacial pain (MFP). The last is the one we seek to explore the etiology of this pain is explained using a biological-psychological model, which reflects the complex interaction between physical factors, behavioral, social and emotional influences (3). The pain may last from weeks to many months; it is usually more severe on one side of the face, especially at pre-auricular area (front ear). Intensity of the pain is usually moderate; it has a squeezing, dull nature. It worsens during mouth opening and often causes opening restriction (5, 4). One can find trigger points where the pain is harsh and radiates to remote areas. Treatment is often integrated, multi-systemic and comprehensive (7, 6): physical therapy, behavioral therapy, night splints, Trigger point injection, and the use of drugs from different families are used to manage and treat MVP. Among the drugs that we use routinely are: Amitriptyline and nortriptyline from the family of tricyclic antidepressants (TAC's). These drugs were originally intended to treat depression and now days there primary use is to treat chronic pain from muscle origin, the use is in low doses of 10-35 mg /d, with no connection to the anti-depressive effect (8,9,10,11). . Gabapentin is gaba-amino buyic acid (GABA) analogue originally developed as an anti-epileptic (12). This drug is also used as a first treatment in neuropathic pain (13). A study published in 2007 by Kimos et al (14) suggested that using gabapentin at higher doses up to 4200 mg per day is a therapeutic option for myofacial pain. The authors prospectively examined the use of gabapentin versus placebo in myofacial pain over 12 weeks in 50 patients, of whom 36 completed the study, the results demonstrated improvement in any parameter. Another study conducted in our department and accepted for publication in journal of orafacail pain & headache examined retrospectively gabapentin Vs amitriptyline with better results for gabapentin in more complex and widely spread disorder. To gabapentin side effect drug interactions profile better than amitriptyline (16). Moreover, gabapentin has no anticholinergic which usually limits the use of amitriptyline. Therefore, gabapentin may be an attractive alternative for the treatment of MFP. Our clinic use gabapentin routinely as second option after lack of response to amitriptyline. The aim of this study is to compare prospectively the efficacy amitriptyline in low doses up to 20 mg to gabapentin at low doses up to 900mg.

Patients over the age of 18 that will come to orofacial pain clinic in the department of Oral medicine, and which will be diagnosed as suffering from facial pain originating from chewing muscles (MVP) for at least three months, will be invited to participate in the study. The examination is the one we use routinely and includes: patient demographics: age, sex, marital status, occupation, and medical history. Pain characteristics includes : Location, duration, intensity (subjective), the nature of the pain, whether pain is prolonged or not, frequency and duration of attacks, disruption of sleep, quality of life and everyday functioning (work, company), whether the pain is accompanied by autonomic of systemic signs and whether the patient suffers from pain in the body outside the region head and neck. Patient will receive a questionnaire examining the accompanying emotional distress (AXIS II). Masticatory muscle involvement will be examined by palpation, load testing, restriction or non-limitation of mouth opening. All of which are routinely use in our department.

Patients will receive an explanation of the nature of the disease and possible treatments. Patients that would like to participate in the study, will sign a consent form, receive a pain questionnaire and start medication treatment which is acceptable in cases of myofacial pain. The drugs that will be used are: amitriptyline up to 20 mg and Gabapentin up to 900 mg. Patients with any side effects will call to receive instructions. After one month, patients will be invited to our clinic. A clinical examination, similar to one mention above will be performed with re-filling of the questionnaires. First medication treatment will discontinue and after two weeks will be replaced with the equivalent drug. Meaning patients that will begin with amitriptyline will continue with gabapentin (after two weeks break) and vice versa (cross over design). After another month patients will be invited to the clinic for further similar clinical examination and questionnaires fulfilling, then, if necessary patients will continue their preferred treatment. . All patients will give their consent to participate in the study.

Criteria for improvement include: 1. Intensity of pain according to VAS scale. 2. The frequency of the attacks. 3. The frequency of use of other drugs (for the treatment of chronic or acute pain). 4. Improving function - open mouth, free jaw movement. 5. Quality Health Index (AXIS II).

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer from chronic pain more than 3 months prior to arrival
* patients who are capable to reach all the visits in the clinic
* Not pregnant women

Exclusion Criteria:

* Patients with other types of non-muscle origin pain
* Patients without a clear diagnosis.
* Patients who are not originally designated to medication treatment (regardless experiment) for various reasons eg pregnancy.
* Patients who are not interested in medication.
* Patients who are not interested or unable to cooperate.
* Patients who suffer from chronic pain less than 3 months prior to arrival
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
pain decrease | 6 weeks
  pain scale measuring

SECONDARY OUTCOMES:
The frequency of use of other drugs | 6 weeks
  breacking drugs registration
Improving function - open mouth, free jaw movement | 6 weeks
  opening mouth measurement

CONTACTS AND LOCATIONS:
Overall Officials: Doron J Aframian, DMD,PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah MO, Jerusalem, Israel

REFERENCES:
- [Background] Tjakkes GH, Reinders JJ, Tenvergert EM, Stegenga B. TMD pain: the effect on health related quality of life and the influence of pain duration. Health Qual Life Outcomes. 2010 May 2;8:46. doi: 10.1186/1477-7525-8-46. PMID 20433769
- [Background] Maixner W, Diatchenko L, Dubner R, Fillingim RB, Greenspan JD, Knott C, Ohrbach R, Weir B, Slade GD. Orofacial pain prospective evaluation and risk assessment study--the OPPERA study. J Pain. 2011 Nov;12(11 Suppl):T4-11.e1-2. doi: 10.1016/j.jpain.2011.08.002. No abstract available. PMID 22074751
- [Background] Benoliel R, Svensson P, Heir GM, Sirois D, Zakrzewska J, Oke-Nwosu J, Torres SR, Greenberg MS, Klasser GD, Katz J, Eliav E. Persistent orofacial muscle pain. Oral Dis. 2011 Apr;17 Suppl 1:23-41. doi: 10.1111/j.1601-0825.2011.01790.x. PMID 21382137
- [Background] Kino K, Sugisaki M, Haketa T, Amemori Y, Ishikawa T, Shibuya T, Sato F, Amagasa T, Shibuya T, Tanabe H, Yoda T, Sakamoto I, Omura K, Miyaoka H. The comparison between pains, difficulties in function, and associating factors of patients in subtypes of temporomandibular disorders. J Oral Rehabil. 2005 May;32(5):315-25. doi: 10.1111/j.1365-2842.2004.01439.x. PMID 15842238
- [Background] Benoliel R, Eliav E, Sharav Y. Classification of chronic orofacial pain: applicability of chronic headache criteria. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Dec;110(6):729-37. doi: 10.1016/j.tripleo.2010.07.009. PMID 21112531
- [Background] Sherman JJ, Turk DC. Nonpharmacologic approaches to the management of myofascial temporomandibular disorders. Curr Pain Headache Rep. 2001 Oct;5(5):421-31. doi: 10.1007/s11916-001-0053-7. PMID 11560807
- [Background] Diamond S, Baltes BJ. Chronic tension headache--treated with amitriptyline--a double-blind study. Headache. 1971 Oct;11(3):110-6. doi: 10.1111/j.1526-4610.1971.hed1103110.x. No abstract available. PMID 4940167
- [Background] Pilowsky I, Hallett EC, Bassett DL, Thomas PG, Penhall RK. A controlled study of amitriptyline in the treatment of chronic pain. Pain. 1982 Oct;14(2):169-179. doi: 10.1016/0304-3959(82)90097-5. PMID 6757842
- [Background] Plesh O, Curtis D, Levine J, McCall WD Jr. Amitriptyline treatment of chronic pain in patients with temporomandibular disorders. J Oral Rehabil. 2000 Oct;27(10):834-41. doi: 10.1046/j.1365-2842.2000.00572.x. PMID 11065017
- [Background] Johannessen SI, Ben-Menachem E. Management of focal-onset seizures: an update on drug treatment. Drugs. 2006;66(13):1701-25. doi: 10.2165/00003495-200666130-00004. PMID 16978035
- [Background] Haviv Y, Zadik Y, Sharav Y, Benoliel R. Painful traumatic trigeminal neuropathy: an open study on the pharmacotherapeutic response to stepped treatment. J Oral Facial Pain Headache. 2014 Winter;28(1):52-60. doi: 10.11607/jop.1154. PMID 24482788
- [Background] Kimos P, Biggs C, Mah J, Heo G, Rashiq S, Thie NM, Major PW. Analgesic action of gabapentin on chronic pain in the masticatory muscles: a randomized controlled trial. Pain. 2007 Jan;127(1-2):151-60. doi: 10.1016/j.pain.2006.08.028. Epub 2006 Oct 9. PMID 17030096
- [Background] Chandra K, Shafiq N, Pandhi P, Gupta S, Malhotra S. Gabapentin versus nortriptyline in post-herpetic neuralgia patients: a randomized, double-blind clinical trial--the GONIP Trial. Int J Clin Pharmacol Ther. 2006 Aug;44(8):358-63. doi: 10.5414/cpp44358. PMID 16961166